CLINICAL TRIAL: NCT03560232
Title: A Randomized Controlled Trial Assessing Noninferiority of Three Antimicrobial Regimens for the Treatment of Grade III Open Fractures
Brief Title: Noninferiority Comparison of Prophylactic Open Fracture Antimicrobial Regimens
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit patients in a timely fashion and unable to recruit sufficient patients
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-028
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Open Fracture; Post-Op Wound Infection
Keywords: Open Fracture; Wound Infection; Antimicrobial Prophylaxis; Cefazolin; Gentamicin; Ceftriaxone; Ampicillin/Sulbactam; Clindamycin; Piperacillin/tazobactam
MeSH Terms: conditions — Fractures, Open; Surgical Wound Infection; Wound Infection | interventions — Ceftriaxone; sultamicillin; Piperacillin, Tazobactam Drug Combination; Cefazolin; Gentamicins; Clindamycin

STUDY DESIGN:
Intervention Model Description: Randomized, open-label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cefazolin + Gentamicin (Active Comparator): [Cefazolin]
  Initial dose:
  * Cefazolin 2g IV x1 dose (patient weight < 120kg)
  * Cefazolin 3g IV x1 dose (patient weight >/= 120kg)
  Subsequent dose:
  * Cefazolin 2g IV every 8 hrs (CrCl >/= 40 mL/min)
  * Cefazolin 2g IV every 12 hrs (CrCl 20-39 mL/min)
  * Cefazolin 2g IV every 24 hrs (CrCl < 20 mL/min)
  Duration:
  * 24 hrs post-op after soft tissue coverage or total of 72 hrs, whichever comes first
  [Gentamicin]
  Initial dose:
  * If Patient age </= 80 years old: 5 mg/kg adjusted body weight x1 dose (Max dose 500 mg)
  * If Patient age >80 years old: 3 mg/kg adjusted body weight x1 dose (Max dose 300 mg)
  Subsequent dose:
  * Pharmacy Consult to dose gentamicin
  Duration:
  * 24 hrs post-op after soft tissue coverage or total of 72 hrs, whichever comes first
  Interventions: Drug: Cefazolin + Gentamicin
- Ceftriaxone (Active Comparator): Initial dose:
  * Ceftriaxone 2g IV x1 dose
  Subsequent dose:
  * Ceftriaxone 2g IV every 24 hours
  Duration:
  * One dose post-op after soft tissue coverage or total of 72 hours, whichever comes first
  Interventions: Drug: Ceftriaxone
- Ampicillin/Sulbactam (Active Comparator): Initial dose:
  * Ampicillin/Sulbactam 3g IV x1 dose
  Subsequent dose:
  * Ampicillin/Sulbactam 3g IV every 6 hours (CrCl >/= 30 mL/min)
  * Ampicillin/Sulbactam 3g IV every 12 hours (CrCl 15-29 mL/min)
  * Ampicillin/Sulbactam 3g IV every 24 hours (CrCl <15 mL/min)
  Duration:
  * 24 hours post-op after soft tissue coverage or total of 72 hours, whichever comes first
  Interventions: Drug: Ampicillin/sulbactam
- Piperacillin/Tazobactam (Active Comparator): Initial dose:
  * Piperacillin/Tazobactam 4.5g IV x1 dose over 30 minutes
  Subsequent dose:
  * Piperacillin/Tazobactam 3.375g IV every 8 hours over 4 hours (CrCl >/= 20 mL/min)
  * Piperacillin/Tazobactam 3.375g IV every 12 hours over 4 hours (CrCl < 20 mL/min)
  Duration:
  * 24 hours post-op after soft tissue coverage or total of 72 hours, whichever comes first
  Interventions: Drug: Piperacillin/tazobactam
- Clindamycin + Gentamicin (Other): Patients with known Penicillin allergy will receive:
  [Clindamycin]
  Initial dose:
  * Clindamycin 900mg IV x1 dose
  Subsequent dose:
  * Clindamycin 600mg IV every 8 hours
  Duration:
  * 24 hours post-op after soft tissue coverage or total of 72 hours, whichever comes first
  [Gentamicin]
  Initial dose:
  * If Patient age </= 80 years old: 5 mg/kg adjusted body weight x1 dose (Max dose 500 mg)
  * If Patient age >80 years old: 3 mg/kg adjusted body weight x1 dose (Max dose 300 mg)
  Subsequent dose:
  * Pharmacy Consult to dose gentamicin
  Duration:
  * 24 hours post-op after soft tissue coverage or total of 72 hours, whichever comes first
  Interventions: Drug: Clindamycin + Gentamicin

INTERVENTIONS:
Drug: Ceftriaxone — See arm description
  Other Names: Rocephin
  Arms: Ceftriaxone
Drug: Ampicillin/sulbactam — See arm description
  Other Names: Unasyn
  Arms: Ampicillin/Sulbactam
Drug: Piperacillin/tazobactam — See arm description
  Other Names: Zosyn
  Arms: Piperacillin/Tazobactam
Drug: Cefazolin + Gentamicin — See arm description
  Other Names: Ancef + Garamycin
  Arms: Cefazolin + Gentamicin
Drug: Clindamycin + Gentamicin — See arm description
  Other Names: Cleocin + Garamycin
  Arms: Clindamycin + Gentamicin

SUMMARY:
To demonstrate noninferiority of three different empiric antimicrobial regimens compared to the traditional antimicrobial regimen for the management of grade III open fractures as well as evaluate outcomes among these groups.

DETAILED DESCRIPTION:
Per the EAST practice management guidelines, an open fracture is defined as one in which the fracture fragments communicate with the environment through a break in the skin. The presence of an open fracture, either isolated or as part of a multiple injury complex, increases the risk of infection and soft tissue complications. Open fractures are further classified into Grade I - Grade III fractures per the Gustilo Classification. Grade III fractures are those with the highest likelihood of contamination and infection with infection rates ranging from 10% to 42%.

EAST guidelines currently recommend systemic gram positive coverage for all open fractures with the addition of gram negative coverage for all Grade III fractures. Antibiotics should be initiated as soon as possible following the injury and should be continued for 72 hours after the injury or not greater than 24 hours after soft tissue coverage was obtained. Traditionally, patients received the combination of Cefazolin and Gentamicin as the preferred prophylactic antibiotic regimen, despite the need for multiple antibiotics and the risk of nephrotoxicity associated with aminoglycosides. Whether there is clinically a more ideal prophylactic antibiotic available remains to be seen. This proposed research initiative is intended to evaluate several antibiotic regimens with similar spectrums of activity to see if there is an equally effective single agent with minimal nephrotoxicity associated with its use. In selecting the study antibiotics to be utilized in the protocol, available information was obtained regarding timing of antibiotics, organisms identified by culture results, and any studies available on specific antibiotic regimens. In regards to timing, there is evidence to support that time to antibiotics and time to the operating room may be more important than the particular antibiotic itself. Additionally, a recent study from 2015 looked at the organisms identified from culture results for Grade I through Grade III fractures in Germany. The vast majority of cultures obtained were gram positive organisms, even in the Grade III fractures, and included Staphylococcus epidermidis, Staphylococcus aureus, Staphylococcus capitis, various Streptococcus species, Enterococcus faecium and Corynebacterium. Interestingly, the only gram negative organism identified in the study was Escherichia coli. Lastly, when trying to identify antibiotic specific studies, a recent study was identified looking at Ceftriaxone as the agent of choice, while limiting the use of vancomycin and aminoglycosides. The conclusion of the study showed a significant decrease in vancomycin and aminoglycosides administered with no increase in infection rates.

Here at St. Elizabeth Youngstown Hospital, the investigator's current trauma and orthopedics practice management guideline has been reviewed and changed multiple times in the past several years. For the vast majority of time, the recommendation has been to use the traditional cefazolin/gentamicin combination. However, several cases of nephrotoxicity led to some hesitation in utilizing this regimen. Therefore, for a short time period, piperacillin/tazobactam was being used for all Grade III fractures instead. At present however, due to conflicting concerns regarding antimicrobial stewardship with utilizing broad spectrum piperacillin/tazobactam with the nephrotoxicity concerns of gentamicin, the approved guideline utilizes cefazolin/gentamicin for patients under 65 years of age and piperacillin/tazobactam for all patients greater than or equal to 65 years of age. This study aims to evaluate non-inferiority of ampicillin/sulbactam, ceftriaxone, and piperacillin/tazobactam when compared to the traditional regimen of cefazolin/gentamicin for grade III open fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age great than/equal to 18 years
* Diagnosis of Grade III open fracture

Exclusion Criteria:

* Water-borne injury
* Farm-related injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Post-surgical site wound infections | 1 year
  The primary outcome for this study is the number of post-surgical site wound infections, defined as initiation of antibiotics for surgical-site infection and/or need for surgical debridement of site. The acceptable infection rate per Trauma Practice Management Guidelines states a rate less than 20%.

SECONDARY OUTCOMES:
Incidence of acute kidney injury | Hospital admission
  Incidence of acute kidney injury during hospital admission will be collected and compared to the other antibiotic regimens.
  Acute kidney injury is defined as (per KDIGO guidelines):
  * An increase in SCr by 0.3 mg/dL within 48 hours OR
  * Increase in SCr to 1.5 times baseline within the previous 7 days OR
  * Urine volume less than 0.5 mL/kg/h for 6 hours
Average cost of antibiotic therapy per patient | Hospital admission
  Cost per patient of each antibiotic therapy will be calculated and compared to the other antibiotic regimens
Time to antibiotic therapy | Hospital admission
  Time from arrival to receiving first dose of antibiotic therapy will be collected (Goal within 30 minutes of arrival).

CONTACTS AND LOCATIONS:
Overall Officials: Natalie I Rine, PharmD, Study Chair — MercyHealth Youngstown; Paul T Miller, PharmD, Study Chair — MercyHealth Youngstown; Tyson T Schrickel, MD, Study Chair — MercyHealth Youngstown; Stuart Drew, DO, Study Chair — MercyHealth Youngstown; David J Gemmel, PhD, Study Chair — MercyHealth Youngstown; Chad W Donley, MD, Principal Investigator — MercyHealth Youngstown; Allison R Lauver, PharmD, Study Chair — MercyHealth Youngstown
Locations (2):
- United States (2):
  - St. Joseph Warren Hospital, Warren, Ohio
  - St. Elizabeth Youngstown Hospital, Youngstown, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gustilo RB, Mendoza RM, Williams DN. Problems in the management of type III (severe) open fractures: a new classification of type III open fractures. J Trauma. 1984 Aug;24(8):742-6. doi: 10.1097/00005373-198408000-00009. PMID 6471139
- [Background] Hoff WS, Bonadies JA, Cachecho R, Dorlac WC. East Practice Management Guidelines Work Group: update to practice management guidelines for prophylactic antibiotic use in open fractures. J Trauma. 2011 Mar;70(3):751-4. doi: 10.1097/TA.0b013e31820930e5. No abstract available. PMID 21610369
- [Background] Lack WD, Karunakar MA, Angerame MR, Seymour RB, Sims S, Kellam JF, Bosse MJ. Type III open tibia fractures: immediate antibiotic prophylaxis minimizes infection. J Orthop Trauma. 2015 Jan;29(1):1-6. doi: 10.1097/BOT.0000000000000262. PMID 25526095
- [Background] Otchwemah R, Grams V, Tjardes T, Shafizadeh S, Bathis H, Maegele M, Messler S, Bouillon B, Probst C. Bacterial contamination of open fractures - pathogens, antibiotic resistances and therapeutic regimes in four hospitals of the trauma network Cologne, Germany. Injury. 2015 Oct;46 Suppl 4:S104-8. doi: 10.1016/S0020-1383(15)30027-9. PMID 26542854
- [Background] Rodriguez L, Jung HS, Goulet JA, Cicalo A, Machado-Aranda DA, Napolitano LM. Evidence-based protocol for prophylactic antibiotics in open fractures: improved antibiotic stewardship with no increase in infection rates. J Trauma Acute Care Surg. 2014 Sep;77(3):400-7; discussion 407-8; quiz 524. doi: 10.1097/TA.0000000000000398. PMID 25159242
- [Background] Lenarz CJ, Watson JT, Moed BR, Israel H, Mullen JD, Macdonald JB. Timing of wound closure in open fractures based on cultures obtained after debridement. J Bone Joint Surg Am. 2010 Aug 18;92(10):1921-6. doi: 10.2106/JBJS.I.00547. Epub 2010 Jul 21. PMID 20660225